CLINICAL TRIAL: NCT04682444
Title: A Prospective Single-blind Comparative Clinical Study of Efficacy and Safety of Amizon 0.25 g Tablets, Manufactured by Farmak JSC, in Patients With ARVI, Including Influenza.
Brief Title: Efficacy and Safety of Enisamium Iodide for the Treatment of Acute Respiratory Viral Infections, Including Influenza.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AM-STP-2-2008
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-11

CONDITIONS: Acute Respiratory Viral Infections; Human Influenza
Keywords: Viral infections; Amizon; Enisamium iodide; Influenza
MeSH Terms: conditions — Influenza, Human; Virus Diseases | interventions — enisamium iodide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor) Matching placebo tablet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Active Treatment - Amizon (Experimental): Patient who were randomized into Group 1 ingested Amizon tablets 500 mg (as 2 tablets, each tablet containing 250 mg enisamium iodide) after a meal, 3 times a day, for 7 days.
  Interventions: Drug: Enisamium Iodide
- Group 2 - Placebo (Placebo Comparator): Patient who were randomized into Group 2 ingested placebo tablets 500 mg (2 tablets), after a meal 3 times a day, for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Enisamium Iodide — Patients ingested Amizon tablets without chewing, after meal, as follows: 2 tablets (total dose 500 mg) 3 times a day, for 7 days. Each tablet contains 250 mg of Nmethyl-4-N-methyl-4-benzylcarbamidopyridinium iodide (INN enisamium iodide).
  Other Names: Amizon
  Arms: Group 1 - Active Treatment - Amizon
Drug: Placebo — Patients ingested placebo tablets without chewing, after meal, in the dose 500 mg (2 tablets), 3 times a day, for 7 days.
  Arms: Group 2 - Placebo

SUMMARY:
This randomized, single blind clinical study was conducted to investigate the clinical efficacy and safety of the drug Amizon (enisamium iodide), in comparison with placebo for the treatment of patients with acute respiratory viral infections (ARVI), including influenza. Enisamium iodide is an antiviral small molecule.

Adult patients were enrolled and randomised into 2 groups. On the first day of the onset of symptoms of ARVI, one group of patients took Amizon tablets (active ingredient enisamium iodide) for 7 days; the other group of patients took matching placebo tablets for 7 days. Examination and observation of all participants was done for up to 14 days after the first intake of the study drug.

The effect of treatment was assessed by subjective reporting of the symptoms of ARVI and influenza, using a predefined symptom scale score system.

Objective assessment was performed by measuring vitals signs, laboratory tests (including blood and urine assessment), as well as evaluating the immune status (including measuring the relative concentration of interferon and immunoglobulins).

DETAILED DESCRIPTION:
Numerous studies have shown that influenza vaccines, prepared against the relevant epidemic seasonal vaccine strains, are an effective remedy in prevention of this mass disease and are able to protect about 80% of otherwise healthy children and adults. However, to develop vaccines against the emerging new pandemic strain of the influenza virus and produce them in the necessary amounts requires at least 6 months. During such interim periods, sufficient protection of the population is essential by effective measures for treatment and prevention of influenza.

This randomized, single-blind, clinical study was conducted to investigate the clinical efficacy and safety of the drug Amizon (N-methyl-4-benzylcarbamidopyridinium iodide, international nonproprietary name enisamium iodide) compared with placebo, for the treatment of patients with ARVI, including influenza.

Enisamium iodide is an antiviral small molecule. Enisamium can directly inhibit influenza viral RNA replication.

The study design was: randomised, single-blind, 2 parallel groups. Adult patients (18-60 y) with symptoms of ARVI, including influenza took either Amizon tablets (active ingredient enisamium iodide) for 7 days; in the control group patients took placebo tablets for 7 days. Study visits occurred on Day 0 (screening, examination, check inclusion/exclusion criteria, enrollment, randomization, and first intake of study drug); further study visits were on Day 3, Day 7, and Day 14.

The effect of treatment was assessed by questioning the patients regarding ARVI and influenza symptoms that included pain, headache, general weakness, sore throat, pain in the joints, fatigue, runny and itchy nose. The severity of symptoms was recorded using a 4-point Likert scale.

Further evaluation of the treatment was performed by measuring the vitals signs, laboratory tests that included blood and urine analysis, biochemical analysis, as well as assessing the immune status (including measuring the absolute lymphocytes count, and evaluating the relative concentration of interferon (IFN)-alpha and IFN-gamma, and immunoglobulin (Ig) A, M, and G (IgA, IgM, and IgG).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 to 60 years
* Patients with ARVI, including influenza, starting not later than for 1 day prior to inclusion in the study:
* The body temperature measured axillary above 37.2 °C
* Presence of one of the signs of respiratory disease (runny nose, cough, pain / tickling in the throat)
* Presence of one of the systemic symptoms (weakness, myalgia, headache , chills, sweating)
* Provide written informed consent
* Ability to understand the nature of the study and provide written informed consent in accordance with Good Clinical Practice (GCP) and local law

Exclusion Criteria:

* Age over 60 years and under 18 years old
* Presence of allergic reactions
* Intolerance to NSAIDs and iodine-containing drugs
* Hypersensitivity to the components of the drug
* Mental illness that impedes compliance with the research procedure
* Pregnancy or breast-feeding
* Presence of acute, clinically significant respiratory and cardio vascular insufficiency, functional disorders of liver, kidney, digestive tract (ulcer disease) determined at physical examination or by laboratory screening tests
* Presence of congenital defects or serious chronic disease of the lungs, kidneys, cardiovascular system, nervous system, metabolic disorders, psychiatric disorders, confirmed by patients history or during initial examination
* The use of preparations of blood cytokine immunoglobulin in for 3 months prior to the study
* Chronic use of alcohol and / or drugs
* Presence or history of cancer diseases, HIV, hepatitis B and C
* Application of immunosuppressive or immunomodulatory drugs for 6-months prior to the study
* Women of child-bearing potential and who do not use acceptable measure of contraception or do not plan to use those throughout the study
* Any clinical condition that, according to the investigator, will not allow to safely carry out the protocol and take the studied drugs without risk to health
* Patients receiving antiviral therapy,
* Participation in other clinical trials at the present time or during the last 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2009-04-13 (Actual); Primary Completion 2010-01-15 (Actual); Study Completion 2010-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ekatarina A. Okhapkina, Principal Investigator — Smorodintsev Research Institute of Influenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Te Velthuis AJW, Zubkova TG, Shaw M, Mehle A, Boltz D, Gmeinwieser N, Stammer H, Milde J, Muller L, Margitich V. Enisamium Reduces Influenza Virus Shedding and Improves Patient Recovery by Inhibiting Viral RNA Polymerase Activity. Antimicrob Agents Chemother. 2021 Mar 18;65(4):e02605-20. doi: 10.1128/AAC.02605-20. Print 2021 Mar 18. PMID 33558285

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 - Active Treatment: Patient who were randomized into Group 1 ingested Amizon tablets 500 mg (2 tablets) after a meal, 3 times a day, for 7 days; each tablet contains 250 mg of enisamium iodide.
  Enisamium Iodide: Patients ingested Amizon tablets without chewing, after meal, as follows: 2 tablets (total dose 500 mg) 3 times a day, for 7 days. Each tablet contains 250 mg of Nmethyl-4-N-methyl-4-benzylcarbamidopyridinium iodide (INN enisamium iodide).
- Group 2 - Placebo: Patient who were randomized into Group 2 ingested placebo tablets after a meal, at the dose 500 mg (2 tablets), 3 times a day, for 7 days.
  Placebo: Patients ingested placebo tablets without chewing, after meal, in the dose 500 mg (2 tablets), 3 times a day, for 7 days.
Period: Overall Study
Arm/Group | Group 1 - Active Treatment | Group 2 - Placebo
Started | 60 | 40
Completed | 60 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with ARVI, including influenza, with disease onset no later than 1 day prior to inclusion to the study. The diagnosis was based on axillary body temperature ≥ 37.2°C, the presence of at least one symptom of respiratory tract infection (rhinitis, pharyngitis, laryngitis, tracheitis, bronchitis, cough), and one general infection symptom (weakness, malaise, myalgia, headache, fever, decreased appetite). The diagnosis was confirmed by viral antigen immunofluorescence testing of nasal swabs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Active Treatment | Group 2 - Placebo | Total
Number analyzed (Participants) | 60 | 40 | 100
Age, Continuous [Mean (Full Range); unit: years] | 37.0 [19 to 59] | 37.6 [19 to 60] | 37.20 [19 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 26 | 64
  Male | 22 | 14 | 36
Region of Enrollment [Number; unit: participants]
  Russia | 60 | 40 | 100
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 24.4 [17.9 to 32.4] | 25.3 [18.5 to 40.8] | 24.7 [17.9 to 40.8]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Number of Participants -- Absence of Objective Symptoms -- Overall
Description: Count of participants WITHOUT objective symptoms -- overall.
  Objective symptoms of acute respiratory viral infection (ARVI), including influenza, were monitored: fever, pharyngeal hyperemia, rhinitis, arterial blood pressure, enlarged lymph nodes, auscultation findings for lung and heart. Clinical improvement was assessed by the investigator, relating to the severity of clinical symptoms of acute respiratory viral infection (ARVI), including influenza.
  A score system used to assess participants' health. A higher score implies worse outcome.
  Objective symptoms scores were: normal or abnormal blood pressure: 0 or 4 score points; lung auscultation: 0 points; vesicular breath sound and wheezing or crepitation 2 or 4 points, respectively; clear and rhythmic heart sounds -- each 0 points; noisy and arrhythmic heart sounds -- each 2 score points.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 - Active Treatment - Amizon: Patient who were randomized into Group 1 ingested Amizon tablets 500 mg (2 tablets) after a meal, 3 times a day, for 7 days; each tablet contains 250 mg of enisamium iodide.
  Enisamium Iodide: Patients ingested Amizon tablets without chewing, after meal, as follows: 2 tablets (total dose 500 mg) 3 times a day, for 7 days. Each tablet contains 250 mg of Nmethyl-4-N-methyl-4-benzylcarbamidopyridinium iodide (INN enisamium iodide).
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: | 0 | 0
  Study Day 3: | 0 | 0
  Study Day 7: | 9 | 4
  Study Day 14: | 44 | 11
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.5547, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p < 0.0001, Fisher Exact

2. Primary Outcome: Efficacy: Number of Participants -- Days Without Routine Activities -- Summary
Description: Count of participants who had days WITHOUT routine activities.
  Disability to perform routine tasks and activities were reported by the participants to the investigator at each study visit.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 - Active Treatment: Patient who were randomized into Group 1 ingested Amizon tablets 0.5 g (2 tablets) after a meal, 3 times a day, for 7 days; each tablet contains 0.25 g of enisamium iodide.
  Enisamium Iodide: Patients ingested Amizon tablets without chewing, after meal, as follows: 2 tablets (total dose 0.5 g) 3 times a day, for 7 days. Each tablet contains 0.25 g of Nmethyl-4-N-methyl-4-benzylcarbamidopyridinium iodide (INN enisamium iodide).
- Group 2 - Placebo: Patient who were randomized into Group 2 ingested placebo tablets after a meal, at the dose 0.5 g (2 tablets), 3 times a day, for 7 days.
  Placebo: Patients ingested placebo tablets without chewing, after meal, in the dose 0.5 g (2 tablets), 3 times a day, for 7 days.
Arm/Group | Group 1 - Active Treatment | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  0 days disability | 26 | 6
  1 day disability | 20 | 10
  2 days disability | 12 | 9
  > 2 days disability | 2 | 15
Statistical Analysis 1: Comparison: Group 1 - Active Treatment vs Group 2 - Placebo; Fisher's exact test was used for testing without adjustment for baseline status; Test type: Superiority; p = 0.0001, Fisher Exact

3. Primary Outcome: Efficacy: Number of Participants -- Viral Antigens -- Overall
Description: Viral antigens that were evaluated: adenovirus, corona virus, influenza A, influenza B, parainfluenza virus, respiratory syncytial virus.
  Virus antigens were isolated from nasal swabs and detected by using validated immunofluorescence staining methods.
  Efficacy assessment was based on the determination of viral antigen on treatment days (Day 3 and Day 7) compared with the baseline (Day 0) in the active treatment group and the placebo group.
  Results represent the count of participants who did NOT have detectable viral antigens.
Time Frame: Day 0 (baseline), 3, 7.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Day 0 Patients who had no detectable viral antigens | 3 | 4
  Day 3 Patients who had no detectable viral antigens: number analyzed (Participants) | 59 | 40
  Day 3 Patients who had no detectable viral antigens | 42 | 10
  Day 7 Patients who had no detectable viral antigens: number analyzed (Participants) | 59 | 40
  Day 7 Patients who had no detectable viral antigens | 59 | 33
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p < 0.0001, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.0013, Fisher Exact

4. Secondary Outcome: Efficacy: Number of Participants -- Absence of Subjective Symptoms -- Overall
Description: Count of participants WITHOUT overall subjective symptoms.
  Subjective symptoms of acute respiratory viral infection (ARVI) including influenza, that were monitored: elevated body temperature, chills, cough, headache, myalgia, sore throat, weakness.
  Evaluate the number of participants in the treatment and the placebo groups without the subjective symptoms from Day 3 after therapy start.
  Clinical improvement was assessed by the investigator, relating to the severity of clinical symptoms of ARVI, including influenza.
  The subjective symptoms were assessed using a 4-point Likert scale, ranging from score 1 (absent symptoms ) to score 4 (severe symptoms).
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 - Active Treatment - Amizon: Patient who were randomized into Group 1 ingested Amizon tablets 0.5 g (2 tablets) after a meal, 3 times a day, for 7 days; each tablet contains 0.25 g of enisamium iodide.
  Enisamium Iodide: Patients ingested Amizon tablets without chewing, after meal, as follows: 2 tablets (total dose 0.5 g) 3 times a day, for 7 days. Each tablet contains 0.25 g of Nmethyl-4-N-methyl-4-benzylcarbamidopyridinium iodide (INN enisamium iodide).
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: | 0 | 0
  Study Day 3: | 0 | 0
  Study Day 7: | 9 | 1
  Study Day 14: | 57 | 18
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.0474, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p < 0.0001, Fisher Exact

5. Secondary Outcome: Efficacy: Subjective Symptom Sum Score (4-point Likert Scale)
Description: Subjective symptom sum score.
  Subjective symptoms of acute respiratory viral infection (ARVI) including influenza, that were monitored: elevated body temperature, chills, cough, headache, myalgia, sore throat, weakness.
  The subjective symptoms were assessed using a 4-point Likert scale for the individual assessment of the severity of the above 7 symptoms, ranging from absent (0), mild (1), moderate (2), or severe (3).
  A higher score implies worse outcome.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Mean (Full Range); unit: score on a 4-point Likert scale
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
score on a 4-point Likert scale
  Study Day 0: | 15.7 [11 to 19] | 15.4 [11 to 18]
  Study Day 3: | 11 [8 to 15] | 11.9 [9 to 17]
  Study Day 7: | 8.4 [7 to 12] | 9.6 [7 to 14]
  Study Day 14: | 7.1 [7 to 10] | 8.0 [7 to 13]
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority — A mixed model repeated measurement was used, which considered baseline, treatment visit*treatment as fixed and patient as random effect; p = 0.0065, MMRM
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p < 0.0001, MMRM — A mixed model repeated measurement was used, which considered baseline, treatment visit*treatment as fixed and patient as random effect
Statistical Analysis 3: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p < 0.0001, MMRM

6. Secondary Outcome: Efficacy: Number of Participants -- Absence of Subjective Symptom -- Chills
Description: Chills.
  Count of participants WITHOUT the subjective symptom: chills.
  Evaluate the number of participants in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  Clinical improvement was assessed by the investigator, relating to the severity of clinical symptoms of acute respiratory viral infection (ARVI), including influenza.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: Chills | 55 | 38
  Study Day 3: Chills | 60 | 40
  Study Day 7: Chills | 60 | 40
  Study Day 14: Chills | 60 | 40

7. Secondary Outcome: Efficacy: Number of Participants -- Absence of Subjective Symptom -- Cough
Description: Cough.
  Count of participants WITHOUT the subjective symptom: cough.
  Evaluate the number of participants in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  Clinical improvement was assessed by the investigator, relating to the severity of clinical symptoms of acute respiratory viral infection (ARVI), including influenza.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: Cough | 1 | 0
  Study Day 3: Cough | 2 | 0
  Study Day 7: Cough | 22 | 3
  Study Day 14: Cough | 57 | 19
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.5152, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.0009, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p < 0.0001, Fisher Exact

8. Secondary Outcome: Efficacy: Number of Participants -- Absence of Subjective Symptom -- Elevated Body Temperature
Description: Count of participants WITHOUT perceived elevated body temperature.
  Evaluate the number of patients in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  Clinical improvement was assessed by the investigator, relating to the severity of clinical symptoms of acute respiratory viral infection (ARVI), including influenza.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: Patients without perceived elevated body temperature | 0 | 0
  Study Day 3: Patients without perceived elevated body temperature | 44 | 23
  Study Day 7: Patients without perceived elevated body temperature | 60 | 37
  Study Day 14: Patients without perceived elevated body temperature | 60 | 39
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.1253, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.0611, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p = 0.4000, Fisher Exact

9. Secondary Outcome: Efficacy: Number of Participants -- Absence of Subjective Symptom -- Sore Throat
Description: Subjective symptoms.
  Count of participants WITHOUT the subjective symptom: sore throat.
  Evaluate the number of patients in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  Clinical improvement was assessed by the investigator, relating to the severity of clinical symptoms of acute respiratory viral infection (ARVI), including influenza.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: Sore throat | 0 | 0
  Study Day 3: Sore throat | 15 | 7
  Study Day 7: Sore throat | 39 | 19
  Study Day 14: Sore throat | 59 | 35
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.4636, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.1000, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p = 0.0363, Fisher Exact

10. Secondary Outcome: Efficacy: Number of Participants -- Absence of Subjective Symptom -- Headache
Description: Subjective symptoms.
  Count of participants WITHOUT the subjective symptom: headache.
  Evaluate the number of patients in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  Clinical improvement was assessed by the investigator, relating to the severity of clinical symptoms of acute respiratory viral infection (ARVI), including influenza.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: Headache | 4 | 6
  Study Day 3: Headache | 29 | 15
  Study Day 7: Headache | 54 | 27
  Study Day 14: Headache | 60 | 37
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.3107, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.0083, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p = 0.0611, Fisher Exact

11. Secondary Outcome: Efficacy: Number of Participants -- Absence of Subjective Symptom -- Myalgia
Description: Myalgia.
  Count of participants WITHOUT the subjective symptom: myalgia.
  Evaluate the number of participants in the active treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  Clinical improvement was assessed by the investigator, relating to the severity of clinical symptoms of acute respiratory viral infection (ARVI), including influenza.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: Myalgia | 28 | 26
  Study Day 3: Myalgia | 59 | 37
  Study Day 7: Myalgia | 60 | 40
  Study Day 14: Myalgia | 60 | 40
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.2988, Fisher Exact

12. Secondary Outcome: Efficacy: Number of Participants -- Absence of Subjective Symptom -- Weakness
Description: Subjective symptoms.
  Count of participants WITHOUT the subjective symptom: weakness.
  Evaluate the number of participants in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  Clinical improvement was assessed by the investigator, relating to the severity of clinical symptoms of acute respiratory viral infection (ARVI), including influenza.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: Weakness | 1 | 0
  Study Day 3: Weakness | 18 | 1
  Study Day 7: Weakness | 41 | 18
  Study Day 14: Weakness | 58 | 33
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.0005, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.0238, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p = 0.0277, Fisher Exact

13. Secondary Outcome: Efficacy: Number of Participants -- Absence of Objective Symptom -- Body Temperature
Description: Efficacy: Count of participants WITHOUT objective symptom: Body temperature.
  Evaluate the number of patients in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  A score system was used to assess patient health, as described under endpoint #1.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0 | 0 | 0
  Study Day 3 | 44 | 23
  Study Day 7 | 60 | 37
  Study Day 14 | 60 | 39
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.1253, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.0611, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p = 0.4000, Fisher Exact

14. Secondary Outcome: Efficacy: Number of Participants -- Objective Symptom: Body Temperature -- Body Temperature Ranges
Description: Body temperature.
  Count of participants in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  Clinical improvement was assessed by the investigator, with respect to the severity of clinical symptoms of acute respiratory viral infection (ARVI), including influenza.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: >38.1 | 1 | 3
  Study Day 0: 37.6-38.0 | 26 | 12
  Study Day 0: 37.1-37.5 | 33 | 25
  Study Day 0: 36.6-37-0 | 0 | 0
  Study Day 3: >38.1 | 0 | 0
  Study Day 3: 37.6-38.0 | 0 | 1
  Study Day 3: 37.1-37.5 | 16 | 16
  Study Day 3: 36.6-37-0 | 44 | 23
  Study Day 7: >38.1 | 0 | 0
  Study Day 7: 37.6-38.0 | 0 | 0
  Study Day 7: 37.1-37.5 | 0 | 3
  Study Day 7: 36.6-37-0 | 60 | 37
  Study Day 14: >38.1 | 0 | 0
  Study Day 14: 37.6-38.0 | 0 | 0
  Study Day 14: 37.1-37.5 | 0 | 1
  Study Day 14: 36.6-37-0 | 60 | 39

15. Secondary Outcome: Efficacy: Number of Participants -- Absence of Objective Symptom -- Lungs Auscultation
Description: Efficacy: Count of participants WITHOUT objective symptom: Lungs auscultation (abnormal breath sounds, detected using a stethoscope).
  Evaluate the number of patients in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start. A score system was used to assess patient health, as described under endpoint #1.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0 | 0 | 1
  Study Day 3 | 0 | 0
  Study Day 7 | 44 | 12
  Study Day 14 | 15 | 5
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p < 0.0001, Fisher Exact

16. Secondary Outcome: Efficacy: Number of Participants -- Absence of Objective Symptom -- Pharyngeal Hyperemia
Description: Efficacy: Number of participants WITHOUT objective Symptom: Pharyngeal Hyperemia.
  Evaluate the number of participants in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start. A score system was used to assess patient health, as described under endpoint #1.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0 | 0 | 0
  Study Day 3 | 5 | 1
  Study Day 7 | 35 | 19
  Study Day 14 | 59 | 33
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.3973, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.3122, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p = 0.0064, Fisher Exact

17. Secondary Outcome: Efficacy Objective Symptom: Number of Participants -- Pharyngeal Hyperemia -- Severity
Description: Pharyngeal hyperemia.
  Count of participants in the treatment and the placebo groups regarding clinical status from Day 3 after therapy start.
  Severity was assessed by the investigator, using a 4-point score scale: 0 = absent; 1 = mild; 2 = moderate; 3 = severe.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Study Day 0: Absent | 0 | 0
  Study Day 0: Mild | 8 | 4
  Study Day 0: Moderate | 51 | 36
  Study Day 0: Severe | 1 | 0
  Study Day 3: Absent | 5 | 1
  Study Day 3: Mild | 44 | 25
  Study Day 3: Moderate | 11 | 14
  Study Day 3: Severe | 0 | 0
  Study Day 7: Absent | 35 | 19
  Study Day 7: Mild | 24 | 19
  Study Day 7: Moderate | 1 | 2
  Study Day 7: Severe | 0 | 0
  Study Day 14: Absent | 59 | 33
  Study Day 14: Mild | 1 | 7
  Study Day 14: Moderate | 0 | 0
  Study Day 14: Severe | 0 | 0

18. Secondary Outcome: Efficacy: Objective Clinical Sum Score
Description: Objective clinical sum score.
  Objective symptoms of acute respiratory viral infection (ARVI), were monitored. For the objective clinical sum score, clinical status was assessed by the investigator, relating to the severity of clinical symptoms of ARVI, including influenza.
  A score system (score points) that was used to assess participants' health, was based on objective symptoms scores, shown below.
  * Blood pressure: normal=0 points; abnormal=4 points.
  * Lung auscultation: vesicular breath sound=0 points; wheezing=2 points; crepitation=4 points.
  * Heart sound; clear heart sounds=0 points; rhythmic heart sounds=0 points; noisy heart sounds=2 points; arrhythmic heart sounds=2 points.
  A higher score implies worse clinical outcome.
Time Frame: Day 0 (baseline), 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Mean (Standard Error); unit: score
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
score
  Study Day 0: | 9.53 (0.09) | 9.65 (0.17)
  Study Day 3: | 7.37 (0.09) | 7.83 (0.15)
  Study Day 7: | 6.02 (0.13) | 6.48 (0.16)
  Study Day 14: | 4.55 (0.12) | 5.60 (0.17)
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.012, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.036, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 14; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Efficacy: Number of Participants -- Viral Antigens -- Baseline Status
Description: Count of randomised participants and their viral antigen types at baseline.
  Viral antigens evaluated: adenovirus, corona virus, influenza A (and subtypes), influenza B, parainfluenza virus, respiratory syncytial virus.
  Virus antigens were isolated from nasal swabs and detected by using validated immunofluorescence staining methods.
Time Frame: Day 0 (baseline).
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  influenza A (H1N1) | 12 | 9
  Influenza A (H3N2) | 14 | 8
  Influenza B | 7 | 5
  Adenovirus (Mono) | 8 | 8
  Influenza A and Adenovirus (Combination of antigens) | 10 | 4
  Parainfluenza (Mono) | 4 | 1
  Respiratory syncytial virus (Mono) | 2 | 1
  Non-differentiated acute respiratory viral infection (ARVI) | 3 | 4

20. Secondary Outcome: Efficacy: Number of Participants -- Viral Antigen -- Influenza Type A
Description: Count of participants who did NOT have a detectable viral antigen -- influenza Type A
  Virus antigen was isolated from nasal swabs and detected by using validated immunofluorescence staining methods.
  Efficacy assessment was the determination of viral antigen on treatment days (Day 3 and Day 7) compared with the baseline (Day 0) in the active treatment group and the placebo group.
Time Frame: Day 0 (baseline), 3, 7.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 26 | 17
Participants
  Day 0 Patients who had no detectable viral antigen | 0 | 0
  Day 3 Patients who had no detectable viral antigen | 20 | 3
  Day 7 Patients who had no detectable viral antigen: number analyzed (Participants) | 25 | 17
  Day 7 Patients who had no detectable viral antigen | 25 | 16
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.0002, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.4048, Fisher Exact

21. Secondary Outcome: Efficacy: Number of Participants -- Viral Antigen -- Influenza Type A or Type B
Description: Viral antigen:
  Count of participants who did NOT have detectable viral antigen -- influenza Type A or Type B.
  Virus antigen was isolated from nasal swabs and detected by using validated immunofluorescence staining methods.
  Efficacy assessment was the determination of viral antigen on treatment days (Day 3 and Day 7) compared with the baseline (Day 0) in the active treatment group and the placebo group.
Time Frame: Day 0 (baseline), 3, 7.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 33 | 22
Participants
  Day 0 Patients who had no detectable viral antigens | 0 | 0
  Day 3 Patients who had no detectable viral antigens | 25 | 5
  Day 7 Patients who had no detectable viral antigens | 32 | 20
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.0002, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.1614, Fisher Exact

22. Secondary Outcome: Efficacy: Number of Participants -- Viral Antigen -- Influenza Type B
Description: Viral antigen:
  Number of participants who did NOT have detectable viral antigen -- influenza Type B.
  Virus antigen was isolated from nasal swabs and detected by using validated immunofluorescence staining methods.
  Efficacy assessment was the determination of viral antigen on treatment days (Day 3 and Day 7) compared with the baseline (Day 0) in the active treatment group and the placebo group.
Time Frame: Day 0 (baseline), 3, 7.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 7 | 5
Participants
  Day 0 Patients who had no detectable viral antigen | 0 | 0
  Day 3 Patients who had no detectable viral antigen | 5 | 2
  Day 7 Patients who had no detectable viral antigen | 7 | 4
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.5581, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.4167, Fisher Exact

23. Secondary Outcome: Efficacy: Number of Participants -- Viral Antigen -- Adenovirus
Description: Viral antigen:
  Count of participants who did NOT have detectable viral antigen -- Adenovirus.
  Virus antigen was isolated from nasal swabs and detected by using validated immunofluorescence staining methods.
  Efficacy assessment was the determination of viral antigen on treatment days (Day 3 and Day 7) compared with the baseline (Day 0) in the active treatment group and the placebo group.
Time Frame: Day 0 (baseline), 3, 7.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 8 | 8
Participants
  Day 0 Patients who had no detectable viral antigen | 0 | 0
  Day 3 Patients who had no detectable viral antigen: number analyzed (Participants) | 7 | 8
  Day 3 Patients who had no detectable viral antigen | 5 | 1
  Day 7 Patients who had no detectable viral antigen | 8 | 5
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.0406, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.2000, Fisher Exact

24. Secondary Outcome: Efficacy: Number of Participants -- Viral Antigen -- Viral Antigen Combination
Description: Viral antigen:
  Count of participants who did NOT have detectable viral antigen -- viral antigen combination.
  Virus antigens were isolated from nasal swabs and detected by using validated immunofluorescence staining methods.
  Efficacy assessment was the determination of viral antigen on treatment days (Day 3 and Day 7) compared with the baseline (Day 0) in the active treatment group and the placebo group.
Time Frame: Day 0 (baseline), 3, 7.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment - Amizon | Group 2 - Placebo
Number analyzed (Participants) | 10 | 4
Participants
  Day 0 Patients who had no detectable viral antigens | 0 | 0
  Day 3 Patients who had no detectable viral antigens | 5 | 0
  Day 7 Patients who had no detectable viral antigens | 10 | 2
Statistical Analysis 1: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 3; Test type: Superiority; p = 0.2208, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment - Amizon vs Group 2 - Placebo; Day 7; Test type: Superiority; p = 0.0659, Fisher Exact

25. Secondary Outcome: Safety - Laboratory Parameters - Immune Status -- Immunoglobulin A, M, G
Description: Assessment of the immune status was performed by evaluating the concentration in blood serum of immunoglobulin A (IgA), immunoglobulin M (IgM), immunoglobulin G (IgG).
  Determination of IgA, IgM, and IgG was performed by turbidimetry.
Time Frame: Day 0 (baseline), 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Mean (Standard Error); unit: grams/liter
Arm/Group | Group 1 - Active Treatment | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
grams/liter
  Day 0, IgA | 2.157 (0.117) | 2.273 (0.140)
  Day 0, IgM | 1.442 (0.093) | 1.338 (0.104)
  Day 0, IgG | 12.247 (0.384) | 11.383 (0.336)
  Day 7, IgA | 2.209 (0.129) | 2.303 (0.136)
  Day 7, IgM | 1.525 (0.112) | 1.315 (0.104)
  Day 7, IgG | 12.175 (0.397) | 11.423 (0.345)
  Day 14, IgA | 2.238 (0.131) | 2.296 (0.136)
  Day 14, IgM | 1.552 (0.113) | 1.400 (0.109)
  Day 14, IgG | 12.388 (0.395) | 11.753 (0.390)

26. Secondary Outcome: Safety - Laboratory Parameters -- Immune Status -- Interferon Alpha (IFN-alpha), Interferon Gamma (IFN-gamma)
Description: Assessment of the immune status was performed by evaluating the concentration in blood serum of IFN-alpha and IFN-gamma.
  Determination of interferon alpha (INF-alpha) and interferon gamma (INF-gamma) in human blood serum was carried out using flow cytometer.
Time Frame: Day 0 (baseline), 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Mean (Standard Error); unit: picograms/mL
Arm/Group | Group 1 - Active Treatment | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
picograms/mL
  Day 0, IFN-alpha | 22.290 (1.264) | 22.541 (1.676)
  Day 0, IFN-gamma | 33.168 (0.912) | 33.008 (1.280)
  Day 7, IFN-alpha | 37.563 (1.308) | 31.768 (1.345)
  Day 7, IFN-gamma | 44.670 (0.765) | 30.478 (0.694)
  Day 14, IFN-alpha | 30.072 (1.123) | 29.388 (1.592)
  Day 14, IFN-gamma | 41.313 (0.770) | 30.393 (0.892)
Statistical Analysis 1: Comparison: Group 1 - Active Treatment vs Group 2 - Placebo; Day 0, IFN-alpha; Test type: Superiority; p = 0.941, Fisher Exact
Statistical Analysis 2: Comparison: Group 1 - Active Treatment vs Group 2 - Placebo; Day 0, IFN-gamma; Test type: Superiority; p = 0.943, Fisher Exact
Statistical Analysis 3: Comparison: Group 1 - Active Treatment vs Group 2 - Placebo; Day 7, IFN-alpha; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: Group 1 - Active Treatment vs Group 2 - Placebo; Day 7, IFN-gamma; Test type: Superiority; p < 0.001, Fisher Exact
Statistical Analysis 5: Comparison: Group 1 - Active Treatment vs Group 2 - Placebo; Day 14, IFN-alpha; Test type: Superiority; p = 0.625, Fisher Exact
Statistical Analysis 6: Comparison: Group 1 - Active Treatment vs Group 2 - Placebo; Day 14, IFN-gamma; Test type: Superiority; p < 0.001, Fisher Exact

27. Secondary Outcome: Evaluation Health Status: Number of Participants -- Overall Treatment Efficacy (Assessment by Investigator and by Patient)
Description: Overall treatment efficacy.
  Evaluate the overall efficacy of the treatment by the investigator and by the participants.
  Results show the number of participants for each assessed category of the health status.
Time Frame: Day 3, 7, 14.
Population: Intention-to-treat. All randomized patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Active Treatment | Group 2 - Placebo
Number analyzed (Participants) | 60 | 40
Participants
  Day 3: Investigator: Complete recovery | 0 | 0
  Day 3: Investigator: Significant improve | 39 | 9
  Day 3: Investigator: Moderate improve | 21 | 28
  Day 3: Investigator: No significant change | 0 | 3
  Day 3: Investigator: Worsened | 0 | 0
  Day 3: Patient: Complete recovery | 0 | 0
  Day 3: Patient: Significant improve | 36 | 6
  Day 3: Patient: Moderate improve | 24 | 31
  Day 3: Patient: No significant change | 0 | 3
  Day 3: Patient: Worsened | 0 | 0
  Day 7: Investigator: Complete recovery | 12 | 0
  Day 7: Investigator: Significant improve | 40 | 30
  Day 7: Investigator: Moderate improve | 7 | 8
  Day 7: Investigator: No significant change | 1 | 2
  Day 7: Investigator: Worsened | 0 | 0
  Day 7: Patient: Complete recovery | 11 | 0
  Day 7: Patient: Significant improve | 42 | 27
  Day 7: Patient: Moderate improve | 6 | 10
  Day 7: Patient: No significant change | 1 | 3
  Day 7: Patient: Worsened | 0 | 0
  Day 14: Investigator: Complete recovery | 56 | 13
  Day 14: Investigator: Significant improve | 4 | 21
  Day 14: Investigator: Moderate improve | 0 | 3
  Day 14: Investigator: No significant change | 0 | 3
  Day 14: Investigator: Worsened | 0 | 0
  Day 14: Patient: Complete recovery | 56 | 13
  Day 14: Patient: Significant improve | 4 | 21
  Day 14: Patient: Moderate improve | 0 | 3
  Day 14: Patient: No significant change | 0 | 3
  Day 14: Patient: Worsened | 0 | 0

ADVERSE EVENTS:
Time Frame: From the study start (Day 0), throughout the study treatment (7 days), and up to the follow-up study visit (Day 14).
Description: Adverse event (AE) was defined as any effect (unfavourable from medical viewpoint) that was experienced by a study subject exposed to the investigational drug, irrespective of its relatedness to study drug.
Arm/Group | Group 1 - Active Treatment | Group 2 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/40
Other Adverse Events (participants affected / at risk) | 4/60 | 3/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Active Treatment (N=60) | Group 2 - Placebo (N=40)
Bitter taste in mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0)
Burning sensation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Allergic rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No